CLINICAL TRIAL: NCT05488496
Title: Testing the Effectiveness of a Nature-based Social Intervention on Loneliness Among Lonely Adults in Barcelona - a Randomized Controlled Trial
Brief Title: Testing a Nature-based Social Intervention on Loneliness: the RECETAS-BCN Trial
Acronym: RECETAS-BCN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vic - Central University of Catalonia (Other)
Collaborators: Barcelona Institute for Global Health (Other); Fundacio Salut i Envelliment UAB (Other); Program on Substance Abuse, Public Health Agency, Government of Catalonia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 945095 BCN
Record Dates: First submitted 2022-07-29; First posted 2022-08-04 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Loneliness
Keywords: social prescription; nature-based therapy; mental health; complex intervention; community-based; wellbeing; prevention; urban health; loneliness
MeSH Terms: conditions — Psychological Well-Being | interventions — Referral and Consultation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): The intervention arm will undergo the following steps:
  1. Groups of 5-15 persons living in the same area. Two trained facilitators support the group dynamics fostering empowerment.
  2. Each participant undergoes a one-to one personalized interview with the facilitator(s) to build the relationship and know participants' expectations and characteristics.
  3. 9 sessions of group-based activities to promote peer support and accessibility and engagement with nature-based activities available in their area according to participant's preferences. A collaborative mapping of nature-based community assets will guide the group to the activities they want to approach and test.
  Interventions: Behavioral: Nature-based social intervention (NBSI), referred as Friends in Nature (FiN)
- Control arm (Active Comparator): The control arm will receive individually usual care (e.g. the existing social prescription as available) and a list of community resources based in nature in the area. Usual care is the appropriate comparison rather than a placebo for complex interventions.
  Interventions: Behavioral: Usual care + menu with nature-based activities

INTERVENTIONS:
Behavioral: Nature-based social intervention (NBSI), referred as Friends in Nature (FiN) — The nature-based social prescribing is a multicomponent complex intervention applied by health or social care professionals as facilitators after a specific training.
  It comprises: a psychosocial component and nature-based activities.
  The psychosocial component is adapted from the group dynamic of "Circle of Friends" methodology focused on loneliness (Jansson A, Pitkälä KH, 2021) adapted to the cultural context of Barcelona and the target population of adults living in urban socio-economic vulnerable areas.
  Nature-based activities are chosen by group participants through a co-created menu comprising all local resources in the area related to nature.
  Specifically, participants start with an individual one-to-one session and then they meet once a week for two hours 10 weeks. Each week, participants decide the nature-based activity they wish to conduct.
  Other Names: Amistat a la natura; Amistad en la naturaleza; Friends in Nature
  Arms: Intervention arm
Behavioral: Usual care + menu with nature-based activities — Social prescribing as existing in usual care plus a written menu with the list of nature-based activities in the area.
  Arms: Control arm

SUMMARY:
RECETAS (Re-imagining Environments for Connection and Engagement: Testing Actions for Social Prescribing in Natural Spaces) is an European project (H2020 No 945095) that aims to reduce loneliness by linking lonely people to nature-based social activities through a group-based intervention.

Background: Loneliness is the perception of feeling alone, even if surrounded by people. Nature-based experiences can facilitate dynamic processes of social interactions and it can reduce feelings of loneliness. RECETAS aims design and test a nature-based social intervention (NBSI) that is group-based and includes access to nature as a main component. The testing will be conducted in six different cities: Barcelona, Helsinki, Prague, Marseille, Cuenca in Ecuador and Melbourne. If successful, this will provide an evidence-based approach for using social prescribing to address loneliness.

Hypothesis: NBSI in vulnerable people suffering from loneliness is more effective than usual social and health care on reducing loneliness at post-intervention (10 weeks), 6- and 12-months follow up.

Objectives: to assess the effectiveness of a 10-week NBSI on loneliness in vulnerable people in the area of Barcelona suffering from it compared to usual social and health care at post-intervention, and at 6-, and 12-months post-randomization. We will also explore the processes and perceived impacts of the intervention.

A pilot study will be conducted (September-December 2022) before the RCT intervention (January 2023) with the aim to explore the feasibility and acceptability of the study procedures, including the primary and secondary outcome measures.

Methods: The study design is a randomized controlled trial (RCT) including a process evaluation based on Medical Health Council guidance, a nested qualitative study and a Health Economics evaluation.

The recruitment will be coordinated and operationalized with Community Development Plans (CDP). Individuals will be recruited from primary care settings, third-sector organizations, community groups, and volunteer organisations who screen for loneliness. A total of 316 participants will be randomly allocated in two arms after the baseline assessment: NBSI treatment and control arms. All of them will be asked to sign the informed consent form.

The intervention model is adapted from the "Circle of Friends" methodology developed by the University of Helsinki (Jansson A, Pitkälä KH, 2021).

DETAILED DESCRIPTION:
RECETAS (Re-imagining Environments for Connection and Engagement: Testing Actions for Social Prescribing in Natural Spaces) is a project that addresses loneliness and the role of nature-based social prescription (NBSP) to reduce it. This project has received funding from the European Union's Horizon 2020 research and innovation under grant agreement No 945094. More information at: https://recetasproject.eu/

Background: Loneliness is the perception of feeling alone, even if surrounded by people. It is a growing public health concern due to its impact on morbidity and mortality, being as dangerous as smoking or obesity: it reduces people's lifespan, and it is associated with chronic diseases as well as mental health symptoms. In Europe, 30 million European adults frequently felt lonely. Social prescription is a non-medical community referral approach to connect individuals with community resources to support wellbeing. Nature-based experiences can facilitate dynamic processes of social interactions and it can reduce feelings of loneliness. We will design and test a nature-based social intervention (NBSI) that is group-based and includes access to nature as a main component. The testing will be conducted in six different cities: Barcelona, Helsinki, Prague, Marseille, Cuenca in Ecuador and Melbourne. If successful, this will provide an evidence-based approach for using social prescribing to address loneliness.

Justification: NBSI in urban areas can improve health and mental well-being and reduce loneliness. Investments in nature-based solutions and green infrastructure can be harnessed for health and wellbeing even in times of health emergencies (covid-19). NBSI offers a novel socio-environmental innovation to reduce loneliness by creating the social infrastructure needed to support social and community cohesion.

Hypothesis: NBSI in vulnerable people suffering from loneliness is more effective than usual social and health care on reducing loneliness at post-intervention (10 weeks), 6- and 12-months follow up.

Objectives: to assess the effectiveness and to explore the processes and perceived impacts of NBSI in vulnerable people suffering from loneliness in the area of Barcelona. The specific objective is to assess the effectiveness of a 10-week NBSI on loneliness in vulnerable people suffering from it compared to usual social and health care at post-intervention, and at 6-, and 12-months post-randomization.

A pilot study will be conducted (September-December 2022) before the RCT intervention (January 2023) with the aim to explore the feasibility and acceptability of the study procedures, including the primary and secondary outcome measures.

Methods: The study design corresponds to a randomized controlled trial (RCT). The RCT will include a process evaluation based on Medical Health Council guidance, a nested qualitative study and a Health Economics evaluation. Therefore, overall, the RCT will use a mixed-method approach collecting quantitative information to assess the main outcomes and qualitative methods to explore lived experiences of participants and professionals. ISGlobal coordinates the overall RECETAS project, UVIC-UCC leads the implementation of the RECETAS-BCN and is responsible for the intervention, assessments, process evaluation and qualitative study. FSIE-UAB is responsible for the recruitment and data analysis. The Public Health Agency of Catalonia is involved and provides support to RECETAS-BCN.

The recruitment will be coordinated and operationalized with Community Development Plans (CDP). Individuals will be recruited from primary care settings, third-sector organizations, community groups, and volunteer organisations who screen for loneliness. A total of 316 participants will be randomly allocated in two arms (158 each): NBSP intervention arm and control arm. All of them will be asked to sign the informed consent form.

Participants are randomly assigned to the intervention or control arm after the baseline assessment.

The intervention is a theory-informed, multicomponent, multi-level, behaviorally based complex intervention that requires a specific training to prepare professionals as facilitators. The intervention model is adapted from the "Circle of Friends" methodology developed by the University of Helsinki by Pitkälä KH et al. It consists in: a) individualized session with facilitators (one-to-one interview), b) group-based program (5-15 people) for 9 sessions, once a week, including nature-based activities in the area chosen by the participants. Control group participants will receive usual care, and a list of nature-based resources available in their area.

ELIGIBILITY:
Inclusion Criteria:

1. To be able to give informed consent in Catalan or Spanish and able to participate to the group dynamics and communicate in at least one of these languages.
2. Aged 18 or over;
3. Currently experiencing loneliness according to the screening question "'Do you suffer from loneliness?" answers "feels lonely 'sometimes, often or always'); can walk to the center independently; able to participate in a group dynamics;
4. Willing to undergo study measurements.

Exclusion Criteria:

1. Unable to go outdoors independently due to poor mobility or severe diseases;
2. Poor hearing or sight in case it prevents them to participate of the group dynamics and activities in the nature;
3. Mild, moderate or severe cognitive decline (test de Pfeiffer >2 fails);
4. Any mental health disorder that might interfere with the group dynamics;
5. Severe disease with poor prognosis < 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
De Jong Gierveld Loneliness Scale 11 item | Post-intervention (10 weeks)
  Loneliness
15D instrument of health-related quality of life - 15D (Sintonen) | Post-intervention (10 weeks)
  Health-related quality of life

SECONDARY OUTCOMES:
De Jong Gierveld Loneliness Scale 11 item | Baseline (before intervention), 6- and 12-months follow up
  Loneliness
15D instrument of health-related quality of life - 15D (Sintonen) | Baseline (before intervention), 6- and 12-months follow up.
  Health-related quality of life
Multidimensional scale of perceived social support (MSPSS) | Baseline (before intervention), Post-intervention (10 weeks), 6- and 12-months follow up
  Perceived Social Support
Pain Brief Inventory | Baseline (before intervention), Post-intervention (10 weeks), 6- and 12-months follow up
  Pain
Perceived Stress Scale (PSS-10) | Baseline (before intervention), Post-intervention (10 weeks), 6- and 12-months follow up
  Stress
EURO-QOL 5D-5L | Baseline (before intervention), Post-intervention (10 weeks), 6- and 12-months follow up
  Quality of Life scale to assess cost-effectiveness
ICEpop CAPability measure for Adults (ICECAP-A) | Baseline (before intervention), Post-intervention (10 weeks), 6- and 12-months follow up
  self-report measure of capability wellbeing for adults
Satisfaction with Life scale (SWLS) | Baseline (before intervention), Post-intervention (10 weeks), 6- and 12-months follow up
  Satisfaction with Life scale as part of Wellbeing scales
Spanish Subjective Happiness Scale | Baseline (before intervention), Post-intervention (10 weeks), 6- and 12-months follow up
  Subjective Happiness Scale as part of Wellbeing scales
Spanish adaptation of the Flourishing Scale Spanish adaptation of the Flourishing Scale | Baseline (before intervention), Post-intervention (10 weeks), 6- and 12-months follow up
  Flourishing Scale as part of Wellbeing scales
Cantril Ladder | Baseline (before intervention), Post-intervention (10 weeks), 6- and 12-months follow up
  Wellbeing assessment
Use of health and social services Use of health and social services retrieved from registers | Baseline (before intervention), Post-intervention (10 weeks), 6- and 12-months follow up
  Retrieved from electronic medical records and self reported
Lubben Social Network Scale-6 | Baseline (before intervention), Post-intervention (10 weeks), 6- and 12-months follow up
  Social interaction
Club/association participation | Baseline (before intervention), Post-intervention (10 weeks), 6- and 12-months follow up
  Social interaction
Questions on distance social relations adapted from adhoc questions asked by K. Pitkala team (Helsinki) | Baseline (before intervention), Post-intervention (10 weeks), 6- and 12-months follow up
  Social interaction
PHQ-9 Patient health questionnaire | Baseline (before intervention), Post-intervention (10 weeks), 6- and 12-months follow up
  Affect/Depression
General anxiety disorder (GADS - 7) | Baseline (before intervention), Post-intervention (10 weeks), 6- and 12-months follow up
  Anxiety
SPANE: Scale of positive and negative experience | Baseline (before intervention), Post-intervention (10 weeks), 6- and 12-months follow up
  Emotions
The 6-item neighborhood attachment scale (NAS) | Baseline (before intervention), Post-intervention (10 weeks), 6- and 12-months follow up
  Neighborhood
Neighborhood aesthetics | Baseline (before intervention), Post-intervention (10 weeks), 6- and 12-months follow up
  Neighborhood
Nature Connection Index (NCI) | Baseline (before intervention), Post-intervention (10 weeks), 6- and 12-months follow up
  Nature dose
The International Physical Activity Questionnaires (IPAQ). | Baseline (before intervention), Post-intervention (10 weeks), 6- and 12-months follow up
  Physical activity
Intrinsic motivation Inventory (IMI) | During intervention (4 week) and Post-Intervention (10 weeks)
  Participants subjective experience related to a target activity
Relatedness to Others in Physical Activity Scale (ROPAS) | During the intervention (4 week), Post-intervention (10 weeks), 6- and 12-months follow up.
  Social support

CONTACTS AND LOCATIONS:
Overall Officials: Jill S Litt, PhD, Principal Investigator — Barcelona Institute for Global Health
Locations (1):
- UVic-UCC, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sachs AL, Maso-Aguado M, Bach A, Opacin N, Hill N, Cattaneo L, Coll-Planas L, Johnson K, Hidalgo L, Daher C, Litt J, Bekessy S. Developing a new tool to capture the nature dose to reduce loneliness and improve quality of life. MethodsX. 2024 Sep 19;13:102969. doi: 10.1016/j.mex.2024.102969. eCollection 2024 Dec. PMID 39385940
- [Background] Vert C, Litt JS, Gascon M, Roque M, Maso-Aguado M, Opacin N, Garcia G, Jansson A, Cattaneo L, Bartova A, Briones-Buixassa L, Carbo A, Rautiainen LJ, Hidalgo L, Sachs A, Domenech S, Blancafort-Alias S, Holmerova I, Pitkala KH, Coll-Planas L. Evaluating the feasibility of "Friends in Nature," a complex nature-based social intervention to address loneliness and quality of life in six cities worldwide. Pilot Feasibility Stud. 2024 Nov 30;10(1):146. doi: 10.1186/s40814-024-01575-4. PMID 39616375
- [Background] Coll-Planas L, Carbo-Cardena A, Jansson A, Dostalova V, Bartova A, Rautiainen L, Kolster A, Maso-Aguado M, Briones-Buixassa L, Blancafort-Alias S, Roque-Figuls M, Sachs AL, Casajuana C, Siebert U, Rochau U, Puntscher S, Holmerova I, Pitkala KH, Litt JS. Nature-based social interventions to address loneliness among vulnerable populations: a common study protocol for three related randomized controlled trials in Barcelona, Helsinki, and Prague within the RECETAS European project. BMC Public Health. 2024 Jan 13;24(1):172. doi: 10.1186/s12889-023-17547-x. PMID 38218784
- [Background] Litt, J. S., Coll-Planas, L., Sachs, A. L., Rochau, U., Jansson, A., Dostálová, V., … Pitkälä, K. H. (2024). Nature-based social interventions for people experiencing loneliness: the rationale and overview of the RECETAS project. Cities & Health, 8(3), 418-431. https://doi.org/10.1080/23748834.2023.2300207
- [Background] Jansson A, Pitkala KH. Editorial: Circle of Friends, an Encouraging Intervention for Alleviating Loneliness. J Nutr Health Aging. 2021;25(6):714-715. doi: 10.1007/s12603-021-1615-5. No abstract available. PMID 34179921
- See also: website of the European Projecte RECETAS — https://recetasproject.eu/